CLINICAL TRIAL: NCT01355627
Title: TachoSil® Versus Current Practice in Dura Sealing Techniques for the Prevention of Post-operative Cerebrospinal Fluid (CSF) Leaks in Patients Undergoing Skull Base Surgery: An Open Label, Randomised, Controlled, Multi-centre, Parallel Group Efficacy and Safety Trial.
Brief Title: TASALL - TachoSil® Against Liquor Leak
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-2402-038-SP
Record Dates: First submitted 2011-05-11; First posted 2011-05-18 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-06

CONDITIONS: Cerebrospinal Fluid Leaks
Keywords: CSF leaks; Skull base surgery; pseudomeningocele; TachoSil®; Prevention; post-operative
MeSH Terms: conditions — Cerebrospinal Fluid Leak | interventions — TachoSil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TachoSil® (Experimental)
  Interventions: Procedure: TachoSil®
- Current practice group (Active Comparator)
  Interventions: Procedure: Current Practice

INTERVENTIONS:
Procedure: TachoSil® — Primary suture must be performed. Duraplasty may be performed at the discretion of the investigator. TachoSil® must be applied under aseptic conditions during the closure of the dura.
  Arms: TachoSil®
Procedure: Current Practice — Primary suture must be performed. Duraplasty may be performed at the discretion of the investigator.
  In addition to primary suture, whatever means of dura closure deemed necessary by the investigator may be used with the exception of TachoSil®.
  Arms: Current practice group

SUMMARY:
The primary objective is to demonstrate superiority of TachoSil® compared to current practice as an adjunct in sealing the dura mater. The efficacy of the dura mater sealing must be evaluated post-operatively. The secondary objective is to evaluate the safety of TachoSil® as an adjunct in sealing the dura mater.

The trial population will consist of 726 randomised (1:1) patients elected for skull base surgery. The trial duration consists of screening, surgery, efficacy follow-up after 7±1 weeks and safety follow-up 28±2 weeks after surgery.

ELIGIBILITY:
Main Inclusion Criteria (Positive response):

• Is the surgical approach/procedure consistent with skull base surgery? I.e. one of the following:

* Lateral approach to the foramen magnum: Far lateral, extreme lateral, anterolateral, posterolateral
* Approach to the jugular foramen: Infratemporal, juxta condylar, transjugular
* Approach to the cerebello pontine (CP) angle and petrous apex retrosigmoid
* Approach to the middle fossa: Subtemporal (+/- petrous apex drilling), pterional approach (any fronto temporal approach +/- orbitozygomatic deposition)
* Approach to the anterior fossa: Subfrontal (uni or bilateral)
* Approach to the midline posterior fossa

Main Exclusion Criteria (Negative response):

* Has the patient been subject to neurosurgery involving opening of the dura mater within the last 3 months?
* Is the patient anticipated to undergo any additional neurosurgery involving opening of the dura mater which may affect the efficacy evaluation (e.g. re-operation or anticipation to undergo several neurosurgeries) before the Efficacy Follow-up Week 7±1 week?
* Is the patient anticipated to undergo any additional neurosurgery involving opening of the dura mater which may affect the safety evaluation (e.g. re-operation or anticipation to undergo several neurosurgeries) before the Safety Follow-up Week 28±2 weeks?
* The surgical approach/procedure is consistent with any transcranial or transfacial or combination of transcranial - transfacial approaches with wide defect in the skull base? I.e. any of the following:

  * Trans basal approach
  * Total petrosectomy
  * Trans facial approach
  * Trans sphenoidal approach
  * Endoscopic procedures
  * Trans oral approach (and any extension: Le Fort, mandibulotomy)
* The surgical approach is consistent with one of the following approaches?

  * Translabyrinthine approach
  * Retrolabyrinthine approach
  * Transcochlear (limited transpetrosal) approach
* Did the arachnoid membrane and the CSF containing system remain intact during surgery?
* Does the patient have more than one dura opening (not including dura openings from extraventricular or lumbar drains)?
* Has TachoSil, fibrin or polymer sealants been used during the current surgery prior to randomization?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed, Study Chair — Clinical Trial Operations
Locations (36):
- Nycomed Investigational Site, Graz, Austria
- Belgium (4):
  - Nycomed Investigational Site, Brussels
  - Nycomed Investigational Site, Genk
  - Nycomed Investigational Site, Leuven
  - Nycomed Investigational Site, Liège
- France (7):
  - Nycomed Investigational Site, Grenoble
  - Nycomed Investigational Site, Le Kremlin-Bicêtre
  - Nycomed Investigational Site, Marseille
  - Nycomed Investigational Site, Nice
  - Nycomed Investigational Site, Paris
  - Nycomed Investigational Site, Strasbourg
  - Nycomed Investigational Site, Toulouse
- Germany (5):
  - Nycomed Investigational Site, Freiburg im Breisgau
  - Nycomed Investigational Site, Halle
  - Nycomed Investigational Site, Homburg
  - Nycomed Investigational Site, München
  - Nycomed Investigational Site, Rostock
- Greece (2):
  - Nycomed Investigational Site, Athens
  - Nycomed Investigational Site, Thessaloniki
- Italy (4):
  - Nycomed Investigational Site, Genova
  - Nycomed Investigational Site, Lecce
  - Nycomed Investigational Site, Palermo
  - Nycomed Investigational Site, Siena
- Nycomed Investigational Site, Dammers, Netherlands
- Poland (2):
  - Nycomed Investigational Site, Gdansk
  - Nycomed Investigational Site, Warsaw
- Nycomed Investigational Site, Moscow, Russia
- Spain (6):
  - Nycomed Investigational Site, Barcelona
  - Nycomed Investigational Site, El Palmar
  - Nycomed Investigational Site, Madrid
  - Nycomed Investigational Site, Majadahonda
  - Nycomed Investigational Site, Málaga
  - Nycomed Investigational Site, Santiago de Compostela
- Sweden (3):
  - Nycomed Investigational Site, Gothenburg
  - Nycomed Investigational Site, Lund
  - Nycomed Investigational Site, Stockholm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at thirty-five Centres in a total of 10 countries: Belgium, France, Germany, Greece, Italy The Netherlands, Poland, Russia, Spain and Sweden from 28 April 2011 to 27 June 2013.
Pre-assignment Details: Participants requiring dura sealing techniques for the prevention of post-operative cerebrospinal fluid (CSF) leaks were enrolled; 726 participants were randomized equally in 1 of 2 treatment groups, TachoSil® or Current practice group.
Groups:
- TachoSil®: Primary suture was performed. Duraplasty could be performed at the discretion of the investigator. TachoSil® was applied under aseptic conditions during the closure of the dura.
- Current Practice Group: Primary suture was performed. Duraplasty could be performed at the discretion of the investigator. In addition to primary suture, whatever means of dura closure treatment, alone or in combination, as deemed necessary by the investigator was used with the exception of TachoSil®.
Period: Overall Study
Arm/Group | TachoSil® | Current Practice Group
Started | 362 | 364
Safety Analysis Set | 362 | 364
Full Analysis Set | 361 (One participant's data for final follow-up is missing, completion status could not be confirmed.) | 365 (One participant randomized to Current Practice actually received TachoSil®.)
Completed | 329 | 326
Not Completed | 33 | 38
Not completed — Request By the Patient to Discontinue | 5 | 7
Not completed — Lost to Follow-up | 8 | 7
Not completed — Fatal Adverse Event | 19 | 23
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Measures were based on the Full Analysis Set that included all enrolled randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | TachoSil® | Current Practice Group | Total
Number analyzed (Participants) | 361 | 365 | 726
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (13.80) | 53.2 (14.22) | 53.1 (14.00)
Age, Customized [Number; unit: participants]
  18-65 years | 288 | 293 | 581
  >65 years | 73 | 72 | 145
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 211 | 444
  Male | 128 | 154 | 282
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 355 | 361 | 716
  Asian | 1 | 0 | 1
  Black or African American | 3 | 2 | 5
  American Indian or Alaska Native | 1 | 1 | 2
  Other | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 55 | 62 | 117
  Non-Hispanic and Non-Latino | 295 | 289 | 584
  Unknown | 11 | 14 | 25
Region of Enrollment [Number; unit: participants]
  Belgium | 87 | 87 | 174
  Germany | 33 | 29 | 62
  Spain | 54 | 54 | 108
  France | 24 | 26 | 50
  Greece | 34 | 38 | 72
  Italy | 14 | 14 | 28
  Netherlands | 3 | 2 | 5
  Poland | 59 | 61 | 120
  Russian Federation | 9 | 8 | 17
  Sweden | 44 | 46 | 90
Height [Mean (Standard Deviation); unit: cm] | 167.4 (9.44) | 168.5 (9.18) | 168.0 (9.32)
Weight [Mean (Standard Deviation); unit: kg] | 73.6 (14.40) | 75.2 (16.79) | 74.4 (15.65)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.20 (4.44) | 26.42 (5.10) | 26.31 (4.79)
Fertility Status [Number; unit: participants]
  Fertile | 74 | 74 | 148
  Post-Menopausal | 140 | 111 | 251
  Surgically Sterile | 19 | 26 | 45
  Not Applicable | 128 | 154 | 282

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Evident Verified Post-Operative Cerebrospinal Fluid Leak or Clinically Evident Pseudomeningocele or Treatment Failure
Description: An assessment was performed daily from randomization to Day of Discharge and at the Efficacy Follow-up visit at week 7 ± 1 week. Clinically evident cerebrospinal fluid leak was confirmed by: 1. Glucose concentration test and/or 2. β-2-transferrin test. A clinically evident pseudomeningocele was considered to be present post-operatively if the following criteria were fulfilled: 1. A subcutaneous, visible/palpable fluctuant fluid accumulation was noted at the site of the surgical incision or adjacent to it; 2. It is suspected the fluid accumulation is cerebrospinal fluid. A treatment failure was defined as application of a new and/or different treatment after application of the study treatment or a third application of (or part of) the selected study treatment on the outside of the dura.
Time Frame: Up to 8 Weeks (7 Weeks ± 1 Week)
Population: Full Analysis Population included all enrolled randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TachoSil® | Current Practice Group
Number analyzed (Participants) | 361 | 365
percentage of participants | 6.9 [4.5 to 10.1] | 8.2 [5.6 to 11.5]
Statistical Analysis 1: Comparison: TachoSil® vs Current Practice Group; Test type: Superiority or Other; p = 0.485, Regression, Logistic; Treatment and pooled centre as covariates; Odds Ratio (OR) = 0.82, Standard Error of Mean 0.23 — < 1 implies a smaller likelihood of a TachoSil treated patient to experience a CSF leak

2. Secondary Outcome: Percentage of Participants With Post-Surgical Non-Clinically Evident Post-Operative Pseudomeningocele
Description: Non-clinically evident pseudomeningocele was defined as a cerebrospinal fluid accumulation found on a postoperative computerized tomography (CT) or magnetic resonance imaging (MRI) scan which fulfilled the following criteria according to the radiologist assessment before Day of Discharge: CT Scan-Fluid accumulation seen as Hypodense signal, MRI Scan-Fluid accumulation seen as Hypointense signal in T1-weighted image and/ OR Fluid accumulation seen as Hyperintense signal in T2-weighted image.
Time Frame: Assessment at least once prior to discharge from neurosurgical ward, with the expected discharge from neurosurgical ward after an average of 10 days (Up to 28 Weeks)
Population: Full Analysis Population included all enrolled randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TachoSil® | Current Practice Group
Number analyzed (Participants) | 361 | 365
percentage of participants | 3.0 [1.5 to 5.4] | 3.0 [1.5 to 5.3]

ADVERSE EVENTS:
Time Frame: Safety data were collected from when the patient signed the Informed Consent Form (ICF) until the Safety Follow-up (Up to 28 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TachoSil® | Current Practice Group
Serious Adverse Events (participants affected / at risk) | 94/362 | 97/364
Other Adverse Events (participants affected / at risk) | 92/362 | 102/364
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TachoSil® (N=362) | Current Practice Group (N=364)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 0
Drug effect decreased (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Spinal pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 4
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 7
Meningitis (Infections and infestations) | 5 | 3
Sepsis (Infections and infestations) | 3 | 5
Septic shock (Infections and infestations) | 2 | 1
Bacterial disease carrier (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 1 | 0
Central nervous system infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subdural empyema (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 1
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 4
Meningitis bacterial (Infections and infestations) | 0 | 3
Meningitis staphylococcal (Infections and infestations) | 0 | 1
Oropharyngitis fungal (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Posterior fossa syndrome (Injury, poisoning and procedural complications) | 1 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 0 | 3
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 2
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Escherichia test positive (Investigations) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 1
Pancreatogenous diabetes (Metabolism and nutrition disorders) | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hydrocephalus (Nervous system disorders) | 10 | 8
Cerebral ischaemia (Nervous system disorders) | 4 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 4 | 4
Brain oedema (Nervous system disorders) | 3 | 1
Facial paresis (Nervous system disorders) | 3 | 1
Brain stem haematoma (Nervous system disorders) | 2 | 0
Cerebellar haematoma (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 2 | 3
Cerebral vasoconstriction (Nervous system disorders) | 2 | 2
Cerebrovascular accident (Nervous system disorders) | 2 | 1
VIIth nerve paralysis (Nervous system disorders) | 2 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Anosmia (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Dementia (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 2
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 3
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 2
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Pneumocephalus (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Quadriparesis (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 2
Subdural hygroma (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Brain stem stroke (Nervous system disorders) | 0 | 1
Bulbar palsy (Nervous system disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 3
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cranial nerve palsies multiple (Nervous system disorders) | 0 | 1
Cranial nerve paralysis (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 2
Hemianopia (Nervous system disorders) | 0 | 1
Hypoglossal nerve paresis (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Artery dissection (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Venous insufficiency (Vascular disorders) | 1 | 0
Air embolism (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TachoSil® (N=362) | Current Practice Group (N=364)
Constipation (Gastrointestinal disorders) | 24 | 12
Nausea (Gastrointestinal disorders) | 19 | 16
Pyrexia (General disorders) | 12 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 23
Pneumocephalus (Nervous system disorders) | 21 | 25
Hypertension (Vascular disorders) | 18 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.